CLINICAL TRIAL: NCT04089280
Title: The Effect of Multi-strain Probiotics on Gastrointestinal Symptoms in Patients With Type 2 Diabetes and Metformin Intolerance. A 32-week Prospective, Single Center, Randomized, Placebo Controlled, Cross-over Clinical Trial.
Brief Title: Probiotics in Metformin Intolerant Patients With Type 2 Diabetes
Acronym: ProGasMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Sanprobi Sp. z o.o., Sp. k., Szczecin, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SilesianMU2
Record Dates: First submitted 2019-08-27; First posted 2019-09-13 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Metformin Adverse Reaction
Keywords: diabetes type 2; probiotics; metformin intolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: prospective, single center , interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sanprobi Barrier-multispecies probiotic (Experimental): A randomized placebo-controlled, parallel-group study, crossover-design. Intervention: Sanprobi Barrier-multispecies probiotic product, 2,5 x10 9 cfu/gram or placebo, cross-over design
  Interventions: Dietary Supplement: Sanprobi Barrier-multispecies probiotic
- carrier material of Sanprobi Barrier-multispecies probiotic (Placebo Comparator): A randomized placebo-controlled, parallel-group study, crossover-design. Intervention: placebo comparator (carrier material of Sanprobi Barrier-multispecies probiotic product , not containing bacterial strains,similar appearance as the probiotic, cross-over design
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Sanprobi Barrier-multispecies probiotic — Multi-strain probiotic Sanprobi Barrier (Bifidobacterium lactis W52, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus lactis W19, Lactobacillus lactis W58, Lactobacillus acidophilus W37, Bifidobacterium bifidum W23, Lactobacillus salivarius W24) or placebo. Patients will be randomized to one of the two products ("A" or "B") each containing probiotic/placebo and administered for 12 weeks. After 12 weeks of supplementation, the probiotic/placebo product "A" or "B" will be discontinued and reintroduced again after next 4 weeks - patients will be switched to the other "A or B" group of probiotic/placebo arm. Patients will be administered with 4 capsules per day for 24 weeks (12 weeks for group A probiotic/placebo and 12 weeks for group B probiotic/placebo allowing 4 weeks washout between the group assignment).
  Arms: Sanprobi Barrier-multispecies probiotic
Other: Placebo Comparator — Carrier material of Sanprobi Barrier-multispecies probiotic product, not containing bacterial strains,similar appearance as the probiotic
  Arms: carrier material of Sanprobi Barrier-multispecies probiotic

SUMMARY:
Metformin, the first-line drug in the treatment of type 2 diabetes (T2DM), may cause dose dependent undesirable side-effects like diarrhea, abdominal pain, nausea or bloating which may affect up to 20 % of patients treated with this drug. The mechanism of the gastrointestinal intolerance in patients treated with metformin is poorly understood. The number of studies on this topic increases and data are mounting that metformin treatment is associated with changes in gut bacterial composition. Among other drugs, metformin also leads to enrichment of short chain fatty acids (SCFAs) producing microbiota which exert positive influence on the human metabolic state.

It has been shown that the therapeutic effect of metformin depends on the microbiota and metformin's main site of action in humans is the intestine. It is also known that patients with T2DM, in general, show evidence of gut dysbiosis followed by alterations of an intestinal barrier leading to an increase in intestinal permeability and elevated inflammatory state.

Therefore, it has been speculated that metformin's versatile effect mediated through the gut microbiota is responsible not only for its therapeutic effect but also for its undesirable digestive symptoms.

Probiotics, defined as "live microorganisms, that when administered in adequate amounts, confer a health benefit on the host", may have the potential to modulate the gut bacterial composition. This is why the investigators hypothesize that it may also reduce the intensity of adverse effects associated with metformin use.

The investigators have chosen Sanprobi Barrier multi-strain formula probiotic because it is identical, in relation to bacterial strains and number, to Ecologic® BARRIER which has been proven in in vitro studies to improve the function of epithelial barrier of the intestine. It was also shown that 12-week administration of strains included in Ecologic® BARRIER in obese postmenopausal women improved intestinal barrier permeability marker (lipopolysaccharide) and cardiometabolic risk factors (waist, fat mass, subcutaneous fat, uric acid, total cholesterol, triglycerides, low-density lipoprotein cholesterol, glucose, insulin, and homeostatic model assessment - insulin resistance (HOMA-IR).

DETAILED DESCRIPTION:
The optimal daily dose of metformin is thought to be 2000 mg, however patients with metformin intolerance cannot reach this target dose. Participate in this study are metformin intolerant. Metformin intolerant patients have been defined as those not able to be treated with the metformin daily dose exceeding 1500 mg due to gastrointestinal upset. Patient's metformin intolerance assessment will be questionnaire based (questionnaire adapted from Laura J. Mc Creight et al.). Patients will fill out questionnaires regarding the gastrointestinal symptoms associated with metformin at a dose they did not tolerate and at a time of reduced daily dose of metformin they do tolerate (patients are accepted to have gastrointestinal symptoms which they accept). Sanprobi Barrier probiotic/placebo will be administrated and the gastrointestinal symptoms will be repeatedly assessed with the use of above mentioned questionnaire at certain time points during the study. Patients will be advice to increase the daily dose of metformin as described below. At certain visits patients will undergo the tests measuring the intestinal permeability (blood and stool zonulin immunoenzymatic tests). Inflammatory state will be assessed by measurement of blood C-reactive protein (CRP) as well as blood and stool calprotectin. Zonulin is an endogenous protease, which concentration provides information about the condition of tight junctions between intestinal cells and has been used a a marker of intestinal permeability. Calprotectin, constitutes up to 60% of soluble cytosolic proteins in human neutrophils. In addition, it occurs in monocytes, macrophages and epithelial cells. Therefore, fecal and serum calprotectin content may be proportional to the number of neutrophils migrating through the gastric and intestinal mucosa and may be associated with inflammatory diseases of the gastrointestinal tract. Calprotectin has been widely used in contemporary clinical practice to monitor inflammation of the gut mucosa. CRP blood concentration is a marker of inflammation. Additionally, fecal samples will be used for microbial analysis (16S ribosomal ribonucleic acid (rRNA) sequencing) and blood samples for oxidative stress parameters, HbA1c, lipogram and alanine aminotransferase activity will be collected. Oxidative stress being a disturbance in oxidative balance, has been associated with type 2 diabetes and linked to adverse health effects, including alterations within the intestinal microbiota and vascular endothelium. Probiotics have already been shown to modify the intestinal microbiota and their usage may exert a beneficial effect on the oxidative stress parameters. This will be a 32 - weeks, prospective, single center, randomized, double-blind, cross-over study consisting of 10 site visits and 4 telephone contacts.

Visit 1. Written informed consent for participation in the study and medical history collection.

Visit 2 - month 0. Randomization visit. (within 3 ± 1 days of the visit 1) Fasting state. Blood pressure, heart rate, body mass index (BMI) measurements, waist-hip ratio (WHR).

Blood collection for zonulin and immunoglobulins against zonulin, calprotectin, CRP, HbA1c, hemoglobin (HGB), red blood cells (RBC), white blood cells (WBC), platelet count (PLT), creatinine, lipogram, alanine aminotransferase (ALT) activity and oxidative stress parameters (antioxidant enzymes: superoxide dismutase (SOD), glutathione peroxidase (GPx); catalase (CAT); glutathione reductase (GR), radical damage indicators of free of lipids and proteins: total oxidation capacity (TOC); concentration of lipid hydroperoxides (LHP); concentration of lipofuscin (LPS) - serum and lysate of erythrocytes; concentration of sulphydryl protein (PSH); malondialdehyde (MDA) concentration - serum and erythrocyte lysate; concentration of reduced glutathione (GSH); non-enzymatic antioxidant system: total antioxidant capacity (TAC) of plasma (total antioxidant status (TAS)) .

Stool collection for microbial analysis, short chain fatty acids, zonulin and calprotectin concentration.

Gastrointestinal symptoms questionnaire administration. Randomization to probiotic/placebo group with the permutation method. Patient will be advised to consume 2 capsules in the morning and 2 capsules in the evening. There will be two groups of probiotic/placebo products namely "A" and "B". Patients who will be randomized to probiotic/ placebo "B" at visit 2 will be switched to probiotic/ placebo "A" at visit 6 and patients who will be randomized to group probiotic/ placebo "A" at visit 2 will be switched to probiotic/ placebo "B" at visit 6. The patient will receive two probiotic/ placebo packs containing 120 capsules each.

Visit 3 - month 1 (4 weeks ± 3 days from the visit 2) Gastrointestinal symptoms questionnaire administration. Return of the empty packages or unused probiotic/placebo issued at the visit 2. The patient will receive two probiotic/ placebo packs containing 120 capsules each.

The current dose of metformin will be increased by 500 mg per day if possible.

Visit 3 A - telephone contact (1 week ± 3 days from the visit 3) Gastrointestinal symptoms will be assessed after increasing the dose of metformin. Decision about the possibility of continuing the increased dose of the drug will be made.

Visit 4 - month 2 (4 weeks ± 3 days from the visit 3) Gastrointestinal symptoms questionnaire administration. Return the empty packages or unused probiotic/placebo issued at the visit 3. The patient will receive two probiotic/ placebo packs containing 120 capsules each. Depending on the patient's clinical symptoms and tolerability of previously increased dose of metformin, increasing the dose of metformin (additional 500 mg/day) will be advised in order to achieve metformin dose of at least 2000 mg. In the case of side-effects from the gastrointestinal system, the dose will be reduced to the dose where there were no symptoms or there were symptoms that patients accepts.

Visit 4 A - Telephone contact (1 week ± 3 days from visit 4) Gastrointestinal symptoms will be assessed after increasing the dose of metformin. Decision about the possibility of continuing the increased dose of the drug will be made.

Visit 5 - month 3 (4 weeks ± 3 days from the the visit 4) Fasting state. Blood pressure, heart rate, BMI measurements, WHR. Blood collection for zonulin and immunoglobulins against zonulin, calprotectin, CRP, HbA1c, HGB, RBC, WBC, PLT, creatinine, lipogram, ALT activity and oxidative stress parameters (SOD, GPx,CAT, GR, TOC, LPS, PSH, MDA, GSH, TAS (TAC).) .

Stool collection for microbial analysis, SCFAs, zonulin and calprotectin concentration.

Gastrointestinal symptoms questionnaire administration. Return the empty packages or unused probiotic/placebo issued at the visit 4. Probiotic / placebo will be discontinued.

Visit 6 - month 4. Cross-over visit. (4 weeks ± 3 days from the visit 5).

Fasting state. Blood pressure, heart rate, BMI measurements, WHR. Blood collection for zonulin and immunoglobulins against zonulin, calprotectin, CRP, HbA1c, HGB, RBC, WBC, PLT, creatinine, lipogram, ALT activity and oxidative stress parameters (SOD, GPx,CAT, GR, TOC, LPS, PSH, MDA, GSH, TAS (TAC).) .

Stool collection for microbial analysis, SCFAs, zonulin and calprotectin concentration.

Gastrointestinal symptoms questionnaire administration. Patient will be cross-over to the different group of probiotic/placebo ("A" or "B" as described on the visit 2) and will be advised to consume 2 capsules in the morning and 2 capsules in the evening.

The patient will receive two probiotic/ placebo packs containing 120 capsules each.

Visit 7 - month 5 (4 weeks ± 3 days from the visit 6) Gastrointestinal symptoms questionnaire administration. Return the empty packages or unused probiotic/placebo issued at the visit 6. The patient will receive two probiotic/ placebo packs containing 120 capsules each.

Depending on the patient's clinical symptoms and tolerability of previously increased dose of metformin, increasing the dose of metformin (additional 500 mg/day) will be advised in order to achieve the metformin dose of at least 2000 mg. In the case of side-effects from the gastrointestinal system, the dose will be reduced to the dose where there were no symptoms or there were symptoms that patients accepts.

Visit 7 A - telephone contact (1 week ± 3 days form the visit 7) Gastrointestinal symptoms will be assessed after increasing the dose of metformin. Decision about the possibility of continuing the increased dose of the drug will be made.

Visit 8 - month 6 (4 weeks ± 3 days from the visit 7) Gastrointestinal symptoms questionnaire administration. Return the empty packages or unused probiotic/placebo issued at the visit 7. The patient will receive two probiotic/ placebo packs containing 120 capsules each.

Depending on the patient's clinical symptoms and tolerability of previously increased dose of metformin, increasing the dose of metformin (additional 500 mg/day) will be advised in order to achieve the metformin dose of at least 2000 mg. In the case of side-effects from the gastrointestinal system, the dose will be reduced to the dose where there were no symptoms or there were symptoms that patients accepts.

Visit 8 A - telephone contact (1 week ± 3 days form the visit 7) Gastrointestinal symptoms will be assessed after increasing the dose of metformin. Decision about the possibility of continuing the increased dose of the drug will be made.

Visit 9 - month 7 (4 weeks ± 3 days from the visit 8) Fasting state. Blood pressure, heart rate, BMI measurements, WHR. Blood collection for zonulin and immunoglobulins against zonulin, calprotectin, CRP, HbA1c, HGB, RBC, WBC, PLT, creatinine, lipogram, ALT activity and oxidative stress parameters (SOD, GPx,CAT, GR, TOC, LPS, PSH, MDA, GSH, TAS (TAC).) .

Stool collection for microbial analysis, SCFAs, zonulin and calprotectin concentration.

Gastrointestinal symptoms questionnaire administration. Return the empty packages or unused probiotic/placebo issued at the visit 8 Probiotic / placebo will be discontinued.

Visit 10 - month 8 (4 weeks ± 3 days from the visit 9) Fasting state. Blood pressure, heart rate, BMI measurements, WHR. Blood collection for zonulin and immunoglobulins against zonulin, calprotectin, CRP, HbA1c, HGB, RBC, WBC, PLT, creatinine, lipogram, ALT activity and oxidative stress parameters (SOD, GPx,CAT, GR, TOC, LPS, PSH, MDA, GSH, TAS (TAC).) .

Stool collection for microbial analysis, SCFAs, zonulin and calprotectin concentration.

Gastrointestinal symptoms questionnaire administration. The patient will finish participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation in the clinical trial
2. Age 18-75 years
3. Type 2 diabetes mellitus diagnosed at minimum 6 months prior to the study
4. Metformin intolerance defined as gastrointestinal adverse effects occurrence at the daily metformin dose higher than 1500 mg assessed by the Questionnaire adapted from Laura J. McCreight et al., which disappeared or decreased to the accepted tolerable level after dose reduction to 1500 mg per day.
5. Metformin treatment in the daily dose not higher than 1500 mg
6. Stable metformin dose in the last 3 months before inclusion to the study

Exclusion Criteria:

1. Estimated Glomerular Filtration Rate (eGFR) < 60 ml /min/ 1.73m2
2. Elevation of ALT and aspartate aminotransferase (AST) activity in the blood serum, three times above the reference value
3. Chronic bowel disease
4. Any other acute or chronic disease that may cause gastrointestinal symptoms
5. Acute or chronic pancreatitis
6. Chronic alcohol consumption >30 g/day for men and > 20 g/day for women
7. Antibiotic therapy in the last 6 months prior to the study
8. Probiotics use in the last 3 months before the study
9. Chronic use of steroid drugs or other immunomodulators
10. Heart failure (New York Heart Association (NYHA) III and IV)
11. Pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse gastrointestinal symptoms related to metformin treatment | 32 weeks
  Questionnaire to Assess Character and Severity of Metformin Intolerance (adapted from Laura J. Mc Creight et al.). The score indicates how the patient tolerates metformin.
  Score interpretation:
  0 - 10 = tolerant (T) 11-20 = mild intolerance (MI) 21-30 = intolerant (I) 31-50 = severely intolerant (SI)

SECONDARY OUTCOMES:
Intestinal barrier permeability and inflammation - zonulin blood concentration | 32 weeks
  blood concentration of zonulin
Intestinal barrier permeability and inflammation - immunoglobulins (IG) against zonulin | 32 weeks
  immunoglobulins against zonulin
Intestinal barrier permeability and inflammation - CRP | 32 weeks
  C-reactive protein
Intestinal barrier permeability and inflammation - stool concentration of zonulin | 32 weeks
  stool concentration of zonulin
Intestinal barrier permeability and inflammation - blood concentration of calprotectin | 32 weeks
  blood concentration of calprotectin
Intestinal barrier permeability and inflammation - stool concentration of calprotectin | 32 weeks
  stool concentration of calprotectin
Faecal microbiota composition | 32 weeks
  16S rRNA sequencing
Short chain fatty acids (SCFAs) | 32 weeks
  assessment of short chain fatty acids in stool (gas chromatography)
Cardiometabolic state - lipid parameters | 32 weeks
  lipid parameters
Cardiometabolic state - Body Mass Index | 32 weeks
  Body Mass Index (BMI)
Cardiometabolic state - blood pressure | 32 weeks
  blood pressure
Cardiometabolic state - heart rate | 32 weeks
  heart rate measurements
Cardiometabolic state - HbA1c | 32 weeks
  blood haemoglobin A1c (HbA1c)
Oxidative stress markers - SOD | 32 weeks
  superoxide dismutase
Oxidative stress markers - GPx | 32 weeks
  glutathione peroxidase
Oxidative stress markers - CAT | 32 weeks
  glutathione catalase
Oxidative stress markers - GR | 32 weeks
  glutathione reductase
Oxidative stress markers - TOC | 32 weeks
  total oxidant capacity
Oxidative stress markers - LHP | 32 weeks
  lipid hydroperoxides
Oxidative stress markers - LPS | 32 weeks
  lipofuscin concentration
Oxidative stress markers - PSH | 32 weeks
  protein sulphydryl concentration
Oxidative stress markers - MDA | 32 weeks
  malondialdehyde concentration
Oxidative stress markers - GSH | 32 weeks
  glutathione concentration
Oxidative stress markers - TAS | 32 weeks
  total antioxidant status

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Nabrdalik, Principal Investigator — Medical University of Silesia
Locations (1):
- Department of Internal Diseases, Diabetology and Nephrology, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rena G, Hardie DG, Pearson ER. The mechanisms of action of metformin. Diabetologia. 2017 Sep;60(9):1577-1585. doi: 10.1007/s00125-017-4342-z. Epub 2017 Aug 3. PMID 28776086
- [Background] Bonnet F, Scheen A. Understanding and overcoming metformin gastrointestinal intolerance. Diabetes Obes Metab. 2017 Apr;19(4):473-481. doi: 10.1111/dom.12854. Epub 2017 Feb 22. PMID 27987248
- [Background] McCreight LJ, Stage TB, Connelly P, Lonergan M, Nielsen F, Prehn C, Adamski J, Brosen K, Pearson ER. Pharmacokinetics of metformin in patients with gastrointestinal intolerance. Diabetes Obes Metab. 2018 Jul;20(7):1593-1601. doi: 10.1111/dom.13264. Epub 2018 Mar 23. PMID 29457876
- [Background] Elbere I, Kalnina I, Silamikelis I, Konrade I, Zaharenko L, Sekace K, Radovica-Spalvina I, Fridmanis D, Gudra D, Pirags V, Klovins J. Association of metformin administration with gut microbiome dysbiosis in healthy volunteers. PLoS One. 2018 Sep 27;13(9):e0204317. doi: 10.1371/journal.pone.0204317. eCollection 2018. PMID 30261008
- [Background] Forslund K, Hildebrand F, Nielsen T, Falony G, Le Chatelier E, Sunagawa S, Prifti E, Vieira-Silva S, Gudmundsdottir V, Pedersen HK, Arumugam M, Kristiansen K, Voigt AY, Vestergaard H, Hercog R, Costea PI, Kultima JR, Li J, Jorgensen T, Levenez F, Dore J; MetaHIT consortium; Nielsen HB, Brunak S, Raes J, Hansen T, Wang J, Ehrlich SD, Bork P, Pedersen O. Disentangling type 2 diabetes and metformin treatment signatures in the human gut microbiota. Nature. 2015 Dec 10;528(7581):262-266. doi: 10.1038/nature15766. Epub 2015 Dec 2. PMID 26633628
- [Background] Bordalo Tonucci L, Dos Santos KM, De Luces Fortes Ferreira CL, Ribeiro SM, De Oliveira LL, Martino HS. Gut microbiota and probiotics: Focus on diabetes mellitus. Crit Rev Food Sci Nutr. 2017 Jul 24;57(11):2296-2309. doi: 10.1080/10408398.2014.934438. PMID 26499995
- [Background] Szulinska M, Loniewski I, van Hemert S, Sobieska M, Bogdanski P. Dose-Dependent Effects of Multispecies Probiotic Supplementation on the Lipopolysaccharide (LPS) Level and Cardiometabolic Profile in Obese Postmenopausal Women: A 12-Week Randomized Clinical Trial. Nutrients. 2018 Jun 15;10(6):773. doi: 10.3390/nu10060773. PMID 29914095
- [Background] de Roos NM, Giezenaar CG, Rovers JM, Witteman BJ, Smits MG, van Hemert S. The effects of the multispecies probiotic mixture Ecologic(R)Barrier on migraine: results of an open-label pilot study. Benef Microbes. 2015;6(5):641-6. doi: 10.3920/BM2015.0003. Epub 2015 Apr 22. PMID 25869282
- [Background] Fasano A. Intestinal permeability and its regulation by zonulin: diagnostic and therapeutic implications. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1096-100. doi: 10.1016/j.cgh.2012.08.012. Epub 2012 Aug 16. PMID 22902773
- [Background] Catalan V, Gomez-Ambrosi J, Rodriguez A, Ramirez B, Rotellar F, Valenti V, Silva C, Gil MJ, Fernandez-Real JM, Salvador J, Fruhbeck G. Increased levels of calprotectin in obesity are related to macrophage content: impact on inflammation and effect of weight loss. Mol Med. 2011;17(11-12):1157-67. doi: 10.2119/molmed.2011.00144. Epub 2011 Jul 5. PMID 21738950
- [Background] Zamani B, Sheikhi A, Namazi N, Larijani B, Azadbakht L. The Effects of Supplementation with Probiotic on Biomarkers of Oxidative Stress in Adult Subjects: a Systematic Review and Meta-analysis of Randomized Trials. Probiotics Antimicrob Proteins. 2020 Mar;12(1):102-111. doi: 10.1007/s12602-018-9500-1. PMID 30666617